CLINICAL TRIAL: NCT01535859
Title: A Randomised Controlled Trial of Cabergoline Prophylaxis for Ovarian Hyperstimulation Syndrome in IVF Cycles and Derivation of Biomarkers for OHSS.
Brief Title: Study of Cabergoline for Prevention of Ovarian Hyperstimulation Syndrome (OHSS) in In Vito Fertilization Cycles and Derivation of OHSS Biomarkers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KNMRCNIG1031; NMRC/NIG/1029/2010 (Other Grant/Funding Number: National Medical Research Council)
Record Dates: First submitted 2012-02-15; First posted 2012-02-20 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-06

CONDITIONS: Ovarian Hyperstimulation Syndrome
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — Cabergoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cabergoline (Experimental)
  Interventions: Drug: Cabergoline
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cabergoline — Cabergoline in 0.5mg tablet. 1 tablet daily for 8 days.
  Other Names: Dostinex
  Arms: Cabergoline
Drug: Placebo — 1 tablet daily for 8 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether cabergoline is effective in reducing the incidence and severity of Ovarian Hyperstimulation Syndrome (OHSS), especially for severe cases; and to derive biomarkers for the risk of developing OHSS.

DETAILED DESCRIPTION:
Severe ovarian hyperstimulation syndrome (OHSS) occurs in up to 2% of in-vitro fertilisation (IVF) cycles, resulting in accumulation of fluid in peritoneal, pleural and pericardial cavities, haemo-concentration with resultant venous thromboembolic phenomena, reduced perfusion of vital organs, renal failure, acute respiratory failure, and even death.

The long term aim is to develop a comprehensive strategy in reducing the incidence and severity of OHSS in in-vitro fertilisation (IVF) cycles. Our short term aim (2-3 years) is to test the ability of the dopamine receptor agonist cabergoline in reducing the incidence and severity of OHSS in high risk women undergoing controlled ovarian hyperstimulation (COH) in fresh IVF cycles through a reduction in vasoactive cytokine levels, specifically in serum vascular-endothelial growth factor (VEGF).

Specifically we will:

1. Conduct a randomised double-blind placebo-controlled trial in women at high risk of developing OHSS during a fresh COH-IVF cycle
2. Investigate the serum and follicular fluid levels for potential biomarkers of OHSS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with more than 20 oocytes collected after COH in both gonadotropin-releasing hormone (GnRH) agonist and antagonist cycles

Exclusion Criteria:

* Patients with allergy to dopamine agonists
* Patients who undergo in-vitro maturation cycles
* Patients where GnRH analogues have been used to trigger oocyte maturation in antagonist cycles

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2012-04; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The development of moderate or severe OHSS necessitating admission for management of OHSS. | Within 2 weeks after hCG trigger

SECONDARY OUTCOMES:
The need for abdominal or pleural tap | Within 3 weeks after hCG trigger
Other complications of OHSS (venous thromboembolism, cardiac failure, renal failure, acute respiratory failure, pulmonary oedema and coma) | Within 3 weeks after hCG trigger
Admission into intensive care | Within 3 weeks after hCG trigger
Examination of potential biomarkers for OHSS | 1-2 years

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Sybille Hendricks, MBBS, MRCOG, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Tang H, Mourad SM, Wang A, Zhai SD, Hart RJ. Dopamine agonists for preventing ovarian hyperstimulation syndrome. Cochrane Database Syst Rev. 2021 Apr 14;4(4):CD008605. doi: 10.1002/14651858.CD008605.pub4. PMID 33851429